CLINICAL TRIAL: NCT03696875
Title: Discharge Planning in Emergency Department to Reduce 30-day Adverse Outcomes for Frail Older Patients With Acute Heart Failure: Design and Rationale of DEED FRAIL-AHF Clinical Trial Study
Brief Title: Discharge Planning in Emergency Department for Frail Older With AHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: F. Javier Martin Sanchez (Other)
Responsible Party: Sponsor-Investigator, F. Javier Martin Sanchez, Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEED FRAIL-AHF
Record Dates: First submitted 2018-09-28; First posted 2018-10-05 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Acute Heart Failure; Frail Elderly Syndrome
Keywords: Discharge Planning; Emergency Department; Heart failure; Older; Frail
MeSH Terms: conditions — Emergencies; Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Phase 1: Matched-pair cluster randomized clinical trial. Phase 2: a quasi-experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multilevel Guided Discharge Planning (Experimental)
  Interventions: Other: Multilevel Guided Discharge Planning
- Standard of care (Active Comparator)
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Multilevel Guided Discharge Planning — Clinical recommendations and resources activations + scheduling of early visit with the specialist + communication with primary care + written instruction sheet to the patient
  Arms: Multilevel Guided Discharge Planning
Other: Standard of care — Standard of care
  Arms: Standard of care

SUMMARY:
Objectives: To demonstrate the efficacy of care transition holistic intervention (Multilevel Guided Discharge Planning, MGDP) in reducing 30-day adverse outcomes among frail older patients with acute heart failure (AHF) discharged from Emergency Departments (EDs) and to validate the results of MGDP in real life.

Method: Investigators will select frail patients ≥70 years with primary diagnosis of AHF discharged from EDs. The intervention will consist of MGDP implementation: 1) checklist that includes clinical recommendations and resources activations; 2) scheduling of early visit with the specialist; 3) communication with primary care; 4) providing a written instruction sheet to patient or caregiver. Phase 1: matched-pair cluster randomized clinical trial. EDs were randomly allocated to intervention (n = 10) or control (n = 10) group. Investigators will compare the outcomes between intervention and control groups. Phase 2: a quasi-experimental study. The 20 EDs will carry out the intervention. Investigators will compare the outcomes between phase 1 and phase 2 of intervention group and between phase 1 and phase 2 of control group. The main outcome is a 30-day composite endpoint (ED revisit or hospital admission for AHF and cardiovascular death) after being discharged.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years.
* Diagnosis of descompensated chronic heart failure.
* Screening for frailty positive (ISAR ≥ 2).
* Planned discharge home from Emergency Department (included observation and short stay unit).
* Written informed consent provided by the patient or proxy.

Exclusion Criteria:

* De novo (new onset) acute heart failure (AHF).
* Severe episode of acute heart failure (≥9th decile of MEESSI-AHF Score).
* Uncorrected clinically significant primary valvular disease.
* Acute coronary syndrome currently or within 30 days prior to enrolment.
* Surgery or implanted device within 30 days prior to enrolment.
* Significant arrhythmias.
* Uncorrected systolic blood pressure < 100 mmHg, O2 saturation baseline < 92%, heart rate < 60 or >110 bpm, serum sodium < 130 mmol/l, serum potassium >5,5 mmol/l or hemoglobin <9 g/dL prior to enrolment.
* Planned treatment with vasoactive therapies, ventricular assist device, heart surgery or transplant within 6 months.
* End stage renal disease.
* Severe disability.
* Difficulty intervention due to significant dementia, active delirium or psychiatric disorder.
* Condition with a life expectancy <1 year.
* Length of stay in Emergency Department ≥96 hours.
* Discharged to facility care.
* Inability of outpatient follow-up.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
30-day emergency revisit or hospital admission for acute heart failure or cardiovascular mortality rate after discharge | at 30 days post-discharge
  The proportion of patients who have emergency revisit or hospital admission for acute heart failure or cardiovascular mortality within 30 days after discharge

SECONDARY OUTCOMES:
All-cause emergency revisit rate | at 30 days post-discharge
  The proportion of patients who have ED revisit for all causes within 30 days after discharge
Acute heart failure emergency revisit rate | at 30 days post-discharge
  The proportion of patients who have ED revisit for acute heart failure within 30 days after discharge
Cardiovascular emergency revisit rate | at 30 days post-discharge
  The proportion of patients who have ED revisit for cardiovascular event within 30 days after discharge
All-cause hospitalisation rate | at 30 days post-discharge
  The proportion of patients who have an hospitalisation for all causes within 30 days after discharge
Acute heart failure hospitalisation rate | at 30 days post-discharge
  The proportion of patients who have hospitalisation for acute heart failure within 30 days after discharge
Cardiovascular hospitalisation rate | at 30 days post-discharge
  The proportion of patients who have hospitalisation for cardiovascular events within 30 days after discharge
All-cause mortality rate | at 30 days post-discharge
  The proportion of patients who have all-cause mortality within 30 days after discharge
Cardiovascular mortality rate | at 30 days post-discharge
  The proportion of patients who have cardiovascular mortality within 30 days after discharge
Free-hospitalization survival | at 30 days post-discharge
  Number of days alive out of the hospital
Functional impairment (assessed by self-reported Barthel index) | Change from baseline to 30 days post-discharge
  Barthel index measures the subject's capacity to perform ten activities of daily living (feeding, bathing, grooming, dressing, bowel and bladder control, toileting, chair transfer, ambulation and stair climbing). The sum score ranges from 0 (totally dependent) to 100 (totally independent).
Pharmacological adherence (assessed by Morisky Medication Adherence Scale) | Within 30 days after discharge
  The four-item MGLS measures pharmacological adherence. The score ranges from 0 (perfect adherence) to 4 (some level of non-adherence).
Satisfaction of patient or caregiver about transition of care (assessed by Care Transitions Measure questionnaire) | Within 30 days after discharge
  CTM questionnaire assesses the quality of care transitions, with lower scores indicating a poorer quality transition, and higher scores indicating a better transition.
Quality of live of patients (assessed by EuroQol-5D) | Within 30 days after discharge
  EQ-5D measures of health-related quality of life. The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain